CLINICAL TRIAL: NCT06285799
Title: A Randomised, Double-blind Study to Determine the Safety and Efficacy of Iron Hydroxide Adipate Tartrate (IHAT) in Iron Deficient Premenopausal Women
Brief Title: Safety and Effectiveness of Iron Hydroxide Adipate Tartrate (IHAT) in Iron Deficient Premenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nemysis Ltd (Industry)
Collaborators: RDC Clinical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IHAT_ID_2024
Record Dates: First submitted 2024-02-19; First posted 2024-02-29 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Iron-deficiency
Keywords: Iron deficiency; Iron hydroxide adipate tartrate (IHAT); Iron supplementation
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies | interventions — locust bean gum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low Dose IHAT (Experimental): IHAT in capsule form and carob flour in capsule form - taken as 1 x 100mg IHAT capsule (equivalent to 30mg iron) in the morning with water and 1 x placebo capsule in the evening with water
  Interventions: Drug: Low Dose IHAT
- High Dose IHAT (Experimental): IHAT in capsule form - taken as 2 capsules (2 x 100mg IHAT, equivalent to 60mg iron total) daily with water (1 capsule in the morning and 1 capsule in the evening)
  Interventions: Drug: High Dose IHAT
- Carob flour (Placebo Comparator): Carob flour in capsule form - taken as 2 capsules daily with water (1 capsule in the morning and 1 capsule in the evening)
  Interventions: Drug: Carob Flour

INTERVENTIONS:
Drug: Low Dose IHAT — Once daily dose of 1 IHAT capsule (100mg IHAT per capsule) and once daily dose of 1 placebo capsule (carob flour)
  Arms: Low Dose IHAT
Drug: High Dose IHAT — Twice daily dose of 1 IHAT capsule (100mg IHAT per capsule)
  Arms: High Dose IHAT
Drug: Carob Flour — Twice daily dose of 1 placebo capsule (carob flour)
  Arms: Carob flour

SUMMARY:
This is a double blind, randomised, placebo-controlled trial to evaluate orally-dosed Iron Hydroxide Adipate Tartrate (IHAT) at 2 different dose levels compared to placebo for increasing serum ferritin levels in iron deficient, but otherwise healthy premenopausal women over 12 weeks.

DETAILED DESCRIPTION:
This is a double blind, randomised, placebo-controlled trial to evaluate orally-dosed Iron Hydroxide Adipate Tartrate (IHAT) at 2 different dose levels compared to placebo for increasing serum ferritin levels in iron deficient, but otherwise healthy premenopausal women over 12 weeks.

IHAT is a novel bioavailable source of iron. It is a tartrate-modified, nanoparticulate ferric oxo-hydroxide with similar functional properties and small primary particle size to the iron form found in the ferritin core (ferrihydrite).

In this trial, subjects will be randomly assigned to receive either (1) IHAT once a day, (2) IHAT twice a day or (3) a placebo daily for 12 weeks. The primary endpoint is the correction of iron deficiency at week 12. Secondary endpoints include iron status, iron deficiency symptoms and gastrointestinal symptoms over the course of the 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy iron deficient premenopausal women, with iron deficiency defined as serum ferritin < 30 ug/L and generally healthy as C-reactive protein < 3mg/L (1)
* Able to provide informed consent
* Agree not to participate in another clinical trial while enrolled in this trial
* Agree not to give blood donations during the study
* Agree not to change current diet (subjects adhering to a vegetarian or vegan diet are allowed to participate) and/or exercise frequency or intensity

Exclusion Criteria:

* Anaemia (as determined from the haematocrit and haemoglobin measures) (2)
* Subjects regularly taking iron specific supplements during or 2 months prior to study commencement (the use of other mineral/vitamin/herbal preparations is allowed but should be recorded) (3)
* Any uncontrolled serious illness (4)
* Previously told they have an iron absorption problem
* Receiving/prescribed coumadin (Warfarin), heparin, dalteparin, enoxaparin or other anticoagulation therapy
* active smokers, nicotine use, alcohol (5) or drug (prescription or illegal substances) abuse
* chronic gastrointestinal disorders
* Pregnant/lactating women or women trying to conceive
* Diagnosed depression or mental disorder that is uncontrolled
* Eating disorders
* BMI > 35 kg/m2
* Allergic to any of the ingredients in active or placebo formula
* Any condition which in the opinion of the investigator makes the participant unsuitable for inclusion
* Participants who have participated in any other clinical trial during past 1 month

Footnotes:

1. A blood test is required prior to enrolment into the study to receive trial product. Participants will be required to attend a local pathology collection centre and have serum ferritin and CRP within the required limits to be considered enrolled in the study and be provided with trial product.
2. Anyone considered to be anaemic will be excluded and directed to their GP. In women, anaemia is defined as any of the following: Haemoglobin < 115 g/L, Haematocrit < 35%.
3. Potential participants that are taking supplements that would result in their exclusion must wait an 8-week washout period prior to commencing the study.
4. An uncontrolled illness is any illness that is currently not being treated with a stable dose of medication or is fluctuating in severity. A serious illness is a condition that carries a risk of mortality, negatively impacts quality of life and daily function and/or is burdensome in symptoms and/ or treatments.
5. Chronic past and/or current alcohol use (>14 alcohol drinks/week).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Percentage of women recovering from iron deficiency at week 12 | week 12
  Percentage of women recovering from iron deficiency at week 12, defined as serum ferritin levels of 30 - 150 ug/L

SECONDARY OUTCOMES:
Time to reach normalisation of ferritin levels | Baseline, week 6 and week 12
  Time to reach normalisation of ferritin levels via blood test results
Change in iron status | Baseline, week 6 and week 12
  Iron status assessed by serum ferritin in ug/L, haemoglobin in g/dL, serum iron in uM and transferrin saturation, defined as serum iron divided by total iron binding capacity and expressed as a percentage
Change in fatigue | Baseline, week 6 and week 12
  Change in fatigue via Fatigue Severity Scale
Incidence and prevalence of gastrointestinal side effects | Baseline, week 1-6 and week 12
  Incidence and prevalence of gastrointestinal side effects via gastrointestinal symptom questionnaire
Iron deficiency symptoms | Baseline, week 6 and week 12
  Iron deficiency symptoms via 36-Item Short Form Survey Instrument (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cristina Comelli, PhD, Study Director — Nemysis Ltd
Locations (1):
- RDC Clinical Pty Ltd, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No